CLINICAL TRIAL: NCT04713956
Title: G-CSF+DAC+BUCY vs. G-CSF+DAC+BF Conditioning Regimen for Patients With RAEB-1, RAEB-2 and AML Secondary to MDS Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: G-CSF+DAC+BUCY vs G-CSF+DAC+BF Conditioning Regimen for RAEB-1,REAB-2 and AML Secondary to MDS Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Guangzhou First People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First People's Hospital of Chenzhou (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAC+BUCY vs DAC+BF-MDS-2021
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Myelodysplastic Syndrome; Allogeneic Hematopoietic Stem Cell Transplantation; Conditioning
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Busulfan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF+DAC+BF (Experimental): For patients with RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo- HSCT, Granulocyte Colony-Stimulating Factor (G-CSF)+Decitabine+BF conditioning regimen was G-CSF 5ug/kg/day on days -17 to -10 (when white blood cell is more than 20G/L, stop using G-CSF), Decitabine 20mg/m2/day on days -14 to -10, Busulfan (BU) 3.2 mg/kg/day on days -6 to -3, Fludarabine (FLU) 30mg/m2/ day on days -7 to -3.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor(G-CSF); Drug: Decitabine (DAC); Drug: Busulfan (BU); Drug: Fludarabine (FLU)
- G-CSF+DAC+BUCY (Active Comparator): For patients with RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo- HSCT, Granulocyte Colony-Stimulating Factor (G-CSF)+Decitabine+BUCY conditioning regimen was G-CSF 5ug/kg/day on days -17 to -10 (when white blood cell is more than 20G/L, stop using G-CSF), Decitabine 20mg/m2/day on days -14 to -10, Busulfan (BU) 3.2 mg/kg/day on days -7 to -4, Cyclophosphamide (CY) 60 mg/kg/day on days -3 to -2.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor(G-CSF); Drug: Decitabine (DAC); Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor(G-CSF) — G-CSF was administered at 5 ug/kg/day on days-17 to -10. When white blood cell is more than 20G/L, stop using G-CSF.
Drug: Decitabine (DAC) — Decitabine was administered at 20mg/m2/day on days -14 to -10.
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4 in G-CSF+DAC+BUCY group, and it was administered at 3.2 mg/kg/day on days -6 to -3 in G-CSF+DAC +BF group .
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.
  Arms: G-CSF+DAC+BUCY
Drug: Fludarabine (FLU) — Fludarabine was administered at 30 mg/m2/day on days -7 to -3.
  Arms: G-CSF+DAC+BF

SUMMARY:
Allo-HSCT is the most effective way to cure MDS and AML secondary to MDS. At present, the best conditioning regimen for MDS and AML secondary to MDS undergoing allo-HSCT remains in discussion. In this prospective study, the safety and efficacy of G-CSF+DAC+BUCY and G-CSF+DAC+BF conditioning regimens in RAEB-1, REAB-2 and AML secondary to MDS undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allo-HSCT is the most effective way to cure MDS and AML secondary to MDS. At present, the best conditioning regimen for MDS and AML secondary to MDS undergoing allo-HSCT remains in discussion. Our previous study has showed that G-CSF+DAC+BUCY conditioning regimen could reduce the relapse and improve the survival compared with BUCY conditioning regimen, while the two conditioning regimens both have high non-relapse mortality (NRM). Several retrospective and prospective studies including ours have demonstrated that BF conditioning regimen has a lower NRM compared with BUCY conditioning regimen, while the relapse and survival are similar in patients undergoing BF and BUCY conditioning regimens. Based on the above, we design the prospective randomized controlled study to evaluate the safety and efficacy of G-CSF+DAC+BUCY and G-CSF+DAC+BF conditioning regimens in RAEB-1, REAB-2 and AML secondary to MDS undergoing allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* RAEB-1, REAB-2 and AML Secondary to MDS undergoing allo-HSCT
* 14-65 years

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality (NRM) | 1 year

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
Disease-free survival (DFS) | 1 year
Relapse rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China